CLINICAL TRIAL: NCT00814164
Title: A Phase II Study Evaluating Mechanisms of Resistance Following Treatment With Clofarabine and Daunorubicin in Newly Diagnosed Adult Acute Myeloid Leukemia Patients > or = to 60 Years Old
Brief Title: Clofarabine and Daunorubicin in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000630678; RPCI-I-132208 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Clofarabine; Daunorubicin; Cytogenetic Analysis; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clorafarbine with daunorubicin (Experimental): Patients receive clofarabine IV over 1 hour on days 1-5 and daunorubicin hydrochloride IV over 5 minutes on days 1, 3, and 5.
  Interventions: Drug: clofarabine; Drug: daunorubicin hydrochloride; Genetic: cytogenetic analysis; Genetic: protein expression analysis; Other: immunologic technique; Other: pharmacological study

INTERVENTIONS:
Drug: clofarabine — IV
Drug: daunorubicin hydrochloride — IV
Genetic: cytogenetic analysis — Correlative study
Genetic: protein expression analysis — Correlative Study
Other: immunologic technique — Correlative Study
Other: pharmacological study — Correlative Study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving clofarabine together with daunorubicin may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving clofarabine together with daunorubicin works in treating older patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Study complete response (CR) and CR without platelet recovery (CRp) following treatment with clofarabine and daunorubicin hydrochloride in older patients with newly diagnosed acute myeloid leukemia.

Secondary

* Study disease-free and overall survival of these patients following treatment with this regimen.
* Compare disease-free and overall survival of patients whose cells do or do not demonstrate apoptosis following treatment with this regimen.

OUTLINE:

* Induction therapy: Patients receive clofarabine IV over 1 hour on days 1-5 and daunorubicin hydrochloride IV over 5 minutes on days 1, 3, and 5. Patients are assessed after induction course 1. Patients with ≥ 5% blasts in bone marrow may receive another course of induction therapy beginning between 28-84 days after initiation of course 1. Patients who achieve complete remission (CR) or CR without platelet recovery (CRp) (after 1 or 2 courses of induction therapy) proceed to consolidation therapy.
* Consolidation therapy: Beginning between 28 -84 days after initiation of last course of induction therapy, patients receive clofarabine IV over 1 hour on days 1-3 and daunorubicin hydrochloride IV over 5 minutes on days 1 and 3. Patients may receive a second course of consolidation therapy beginning between 28-84 days of consolidation course 1.

Blood and bone marrow samples are collected periodically to assess response and for pharmacokinetic, cytogenetic, immunophenotyping, and molecular analyses.

After completion of study treatment, patients are followed for at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia

  * At least 10% blasts in the peripheral blood
* De novo or secondary disease
* No acute promyelocytic leukemia with t[15;17] or any other variant
* No clinical evidence of CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* LVEF ≥ 45%
* Estimated glomerular filtration rate ≥ 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for at least 6 months following study treatment
* No known HIV positivity
* Able to comply with study procedures and follow-up examinations
* No psychiatric disorders that would interfere with consent, study participation, or follow-up
* No uncontrolled systemic fungal, bacterial, viral, or other infection (i.e., exhibiting ongoing signs/symptoms related to the infection and without improvement despite appropriate antibiotics or other treatment)
* No history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo induction therapy with both agents
* No other malignancy, unless disease-free for at least 3 years following curative intent therapy

  * Nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are allowed if definitive treatment for the condition has been completed
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* No other severe concurrent disease

PRIOR CONCURRENT THERAPY:

* No other concurrent systemic antileukemic therapy (standard or investigational)
* No concurrent cytotoxic therapy or investigational therapy
* No concurrent alternative medications (e.g., herbal or botanical for anticancer purposes)
* No prior chemotherapy

  * Prior hydroxyurea allowed

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clorafarbine With Daunorubicin
Started | 21
Completed | 2
Not Completed | 19
Not completed — Progression | 7
Not completed — not stated | 7
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: Complete Response/Remission (CR) was defined on morphologic criteria at a single response assessment as follows: A bone marrow aspirate or biopsy of < 5% blasts, with evidence of normal hematopoiesis; Absence of Auer rods in the blast that are present; Absence of extramedullary disease [imaging required only if obtained pretreatment for known site(s) of disease]; If applicable and available, absence of a unique phenotype determined at the pretreatment specimen, as assessed by immunophenotyping; Recovery of peripheral counts (platelets ≥100x109/L, and ANC ≥1.0x109/L). Peripheral count recovery must be documented no earlier than 7 days prior to, and no later than 14 days following, the bone marrow assessment that provides evidence of the CR. Complete Response/Remission without platelet recovery (CRp) was defined as all criteria for CR except for thrombocytopenia (platelet count ≥75x109/L).
Time Frame: 2 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 21
percentage of participant | 38.1 [20.8 to 59.1]

2. Secondary Outcome: Disease-free Survival
Description: Disease-free survival was defined as time from first objective documentation of CR or CRp until the date of first objective documentation of disease relapse or death due to any cause, whichever occurs first.
Time Frame: 5 years
Population: All treated and eligible patients who had first objective documentation of CR or CRp.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 8
months | 6.8 [1.1 to 36.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from date of treatment initiation until date of death due to any cause.
Time Frame: 4 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 21
months | 11.2 [4.2 to 14.2]

4. Secondary Outcome: Differences in Disease-free and Overall Survival Between Patients Whose Cells do or do Not Demonstrate Apoptosis Following Clofarabine and Daunorubicin Hydrochloride Therapy
Time Frame: 4 years
Population: Due to the study's early termination and sponsor's withdrawal of support, data were not collected for this assessment.
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 0

5. Secondary Outcome: Difference in Disease-free and Overall Survival According to p53R2 Protein Sizes
Time Frame: 4 years
Population: Due to the study's early termination and sponsor's withdrawal of support, data were not collected for this assessment.
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 0

6. Secondary Outcome: Difference in Disease-free and Overall Survival According to Multi-drug Resistance Protein Expression
Time Frame: 4 years
Population: Due to the study's early termination and sponsor's withdrawal of support, data were not collected for this assessment.
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 0

7. Secondary Outcome: Difference in Disease-free and Overall Survival Based on Clofarabine Triphosphate Levels
Time Frame: 4 years
Population: Due to the study's early termination and sponsor's withdrawal of support, data were not collected for this assessment.
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 0

8. Secondary Outcome: A Preliminary Relationship Between Treatment Outcome and Biologic Parameters
Time Frame: 4 years
Population: Due to the study's early termination and sponsor's withdrawal of support, data were not collected for this assessment.
Arm/Group | Clorafarbine With Daunorubicin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Clorafarbine With Daunorubicin
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clorafarbine With Daunorubicin (N=21)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Multi-organ failure (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clorafarbine With Daunorubicin (N=21)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Haematotympanum (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Ocular icterus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 16 (20)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Lip dry (Gastrointestinal disorders) | 3 (3)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (14)
Proctitis (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9)
Asthenia (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Infusion site haemorrhage (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 7 (8)
Oedema peripheral (General disorders) | 11 (12)
Pain (General disorders) | 5 (5)
Pneumatosis (General disorders) | 2 (2)
Pyrexia (General disorders) | 9 (11)
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 (10)
Hypersensitivity (Immune system disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 4 (4)
Candidiasis (Infections and infestations) | 4 (5)
Cellulitis (Infections and infestations) | 4 (4)
Cellulitis orbital (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (3)
Infection in an immunocompromised host (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Prothrombin time prolonged (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Lethargy (Nervous system disorders) | 5 (5)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5)
Confusional state (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8)
Mental status changes (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 6 (6)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal mass (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 (5)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 3 (3)
Haemorrhage (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 3 (5)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Pallor (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes